CLINICAL TRIAL: NCT01226251
Title: New "in Vitro" Diagnostic Test for Oral Malodour: First Prototype Evaluation
Brief Title: New "in Vitro" Diagnostic Test for Oral Malodour
Acronym: Striptest
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Gaba International AG (Industry)
Responsible Party: Principal Investigator, Marc Quirynen, PhD DDS, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: 20100914
Record Dates: First submitted 2010-10-12; First posted 2010-10-22 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Halitosis
Keywords: oral malodour; halitosis; Subjects consulting a bad breath clinic
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy adults: Subjects consulting a bad breath clinic at the Department of Periodontology, KULeuven
  Interventions: Device: In vitro chair side test

INTERVENTIONS:
Device: In vitro chair side test — Colour evaluation of a strip
  Other Names: Strip tes for oral malodour GABA (still confidential)

SUMMARY:
This study will assess the ability of a first prototype (strip) of a new chair side test to detect oral malodour. The strip is based on a new enzymatic reaction able to detect amines in saliva. Previous studies already showed significant correlations between oral malodor and the levels of amines in saliva. The limitation in their use as markers of oral malodour is the fact that the detection is usually carried out by complex techniques (High Performance Liquid Chromatography(HPLC)and Solid-Phase Micro Extraction-Gas Chromatography/Mass Spectrometry (SPME-GC/MS)). The results of the new enzymatic reaction can be evaluated by means of a colorimetric scale without necessity of extra apparatus.

The study will be carried out with volunteers recruited at a multidisciplinary consultation for bad breath, organized at the University Hospital Leuven, Belgium.

The paper strip will be used before the routine evaluation (organoleptic score (OS), the gold standard method for the diagnosis of halitosis and the level of volatile sulphur compounds (VSC), the most used adjunct tool to diagnose halitosis).

The results of the new chair side test (strip) will be correlated with the OS and VSC measurements (OralChroma™, Halimeter®). The sensitivity, specificity and positive and negative predicted values of the new chair side test will be calculated. The cut-off values for a yes/no test will be determined. The meaning of color scores will be analyzed to assign a meaningful outcome to each score with relation to odor intensity.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years
* With no evidence of bad breath or bad breath of intra-oral cause (oral malodour)
* Non-smokers or smokers from whom the organoleptic evaluation can be performed (no interference from smoke odour)

Exclusion Criteria:

* Smokers from whom the organoleptic evaluation can not be performed because of interference from smoke odour
* Presence of active caries
* Presence of sinusitis or any other Oro-pharyngeal problem
* On medications which can cause malodour
* Reduced salivary flow due to pathological reasons (e.g. Sjögren syndrome)
* Any oral pathophysiological condition or any oral disease (e.g. oral cancer, mucositis)
* Pregnancy and nursing
* Situation considered not compatible with the study according to the investigator's opinion; the latter includes: persons under homeopathic therapy, patients who used antibiotics during the 2 months before the study, patients frequently using chewing gum, patients under corticosteroids or other serious medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hundred consecutive adult subjects consulting the bad breath clinic who meet the inclusion criteria.
  Number of volunteers extended to 150 in March 2012 (Amendment Research Agreement)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Colour evaluation of the new chair side test | Once (during the first consult to the clinic)
  The colour will be assessed before all the other test and after 4 minutes of contact between the strip and the saliva of the volunteer.

SECONDARY OUTCOMES:
Organoleptic evaluation (OS) | Once (during the first consult to the clinic)
  The OS will be determined by a trained and calibrated judge as described in the literature. Briefly, patients will be asked to count from one to eleven and the judge rated the exhaled air on a 0 to 5 score ( 0 represents absence of odour, 1 is given for barely noticeable odour, 2 for slight malodor, 3 for moderate malodor, 4 for strong malodor and 5 for severe malodor). The judge will also evaluate nasal breath in order to exclude extra-oral causes of halitosis and the odor of a sample of the tongue coating, if present.
Total VSC reading | Once (during the first consult to the clinic)
  The global concentration of sulphur containing compounds will be measured using a portable breath analyzer (Halimeter®, Interscan cooperation, Chatsworth, US. The maximum level attained (ppb) is determined by direct readings from the analog scale of the monitor.
Specific VSC readings | Once (during the first consult to the clinic)
  Hydrogen sulphide, methyl mercaptan and dimethyl sulphide will be measured using a commercially available system (OralChroma™, Abilit Corporation; Osaka City, Japan). This portable gas chromatograph is equipped with an indium oxide semiconductor gas sensor. The concentration values (ppbv) of the three gases will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Quirynen, PhD, DDS, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Department of Periodontology, Faculty of Dentistry, Catholic University of Leuven, Leuven, Belgium